CLINICAL TRIAL: NCT02647983
Title: Multiparametric MRI for Prostate Cancer Localization and Characterization Using Hyperpolarized Pyruvate (13C) Injection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 242-2014
Record Dates: First submitted 2015-12-03; First posted 2016-01-06 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperpolarized Pyruvate (13C) Injection (Experimental): Hyperpolarized Pyruvate (13C) Injection to be used a MRI contrast agent.
  Interventions: Drug: Hyperpolarized Pyruvate (13C) Injection

INTERVENTIONS:
Drug: Hyperpolarized Pyruvate (13C) Injection — Hyperpolarized Pyruvate (13C) Injection is a MRI contrast agent.

SUMMARY:
Prostate cancer is the most common malignancy among men in the United States and Canada. Suspicion of prostate cancer with modern screening tests, such as digital rectal exam (DRE) and prostate serum antigen (PSA) require ultrasound-guided biopsy for pathological diagnosis. However, this technique misses cancer in nearly one quarter of patients and finds clinically insignificant disease in another third of patients, resulting in over-treatment and unnecessary morbidity.

MRI is the best imaging method for prostate cancer detection, but current techniques cannot reliably predict tumour grade and are often unreliable for localizing cancer, particularly within the transition zone, where specificity is low. The primary objective of this pilot study is to evaluate the added benefit of localizing prostate cancer and predicting tumour grade with Hyperpolarized 13C MRI, in addition to traditional T2-weighted and diffusion-weighted MR imaging.

The investigators propose a pilot study, in men diagnosed with prostate cancer awaiting prostatectomy, with the specific goals of comparing pre-operative imaging findings to ground truth histology, using whole-mount prostate specimens. The results of this study will provide insight into the prostate cancer disease signatures with MRI and determine if there is added benefit for incorporation of this new technique into future clinical MRI protocols. If future imaging tests could determine the size, grade and extent of disease, this would open the door for less invasive, localized treatment options with reduced morbidity.

DETAILED DESCRIPTION:
The metabolism of 13C (non-radioactive) enriched pyruvate can be imaged by magnetic resonance (MR) spectroscopy when the nuclear spin of 13C is hyperpolarization enhanced. This technique allows in-vivo separation of [1-13C]pyruvate, [1-13C]lactate, [1-13C]alanine and [13C]bicarbonate signals following intravenous administration of Hyperpolarized Pyruvate (13C) Injection. The total 13C-signal detected in a given tissue depends on the dose administered and distribution to the tissue. The formation rate and relative levels of the metabolites depend on the metabolic needs of the specific tissue. Pre-clinical data indicate that some tumours show substantially higher levels and different ratios of specific metabolites when compared to corresponding normal tissue.

Soon after being taken up by cells within the prostate, [1-13C]pyruvate will be metabolized into various metabolites, including [1-13C]alanine and [13C]bicarbonate (via aerobic metabolism) and [1-13C]lactate (via anaerobic metabolism). It is expected that [1-13C]lactate will be formed in much higher amounts in malignant tissue, where the level of glycolysis is higher than in normal, BPH or inflamed tissues. Therefore, spectroscopic MR imaging of the prostate after administration of Hyperpolarized Pyruvate (13C) Injection, is expected to provide a robust, minimally invasive method to assist in detecting and characterizing prostate cancer, thereby determining which patients should receive further treatment and which should continue to be monitored via routine PSA and DRE testing.

This is a pilot prospective, single-institution study in men with biopsy-proven carcinoma of the prostate. Patient screening and accrual will be completed by a treating Urologist, Radiologist, or study nurse/coordinator. Clinical procedures will be completed at Sunnybrook Health Sciences Centre (SHSC). Eligible subjects will be undergoing radical prostatectomy at SHSC for biopsy-proven T1C disease (cancer found by elevated PSA and needle biopsy only) and serum PSA < 10. For the purpose of analysis, subjects will be divided into three groups based on the grade of cancer found on needle biopsy. A typical subject will be 50-80 years old. The length of this study for participants is approximately 1 hour of scan time.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count (ANC) ≥1500 cells/µl
* Hemoglobin ≥9.0 gm/dL
* Platelets ≥100,000 cells/µL
* Estimated creatinine clearance* ≥60 mL/min

  * by the Cockcroft Gault equation
* Bilirubin within normal range
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within normal range
* Negative test for hepatitis B and hepatitis C
* Eastern Cooperative Oncology Group Status of 0 or 1

Exclusion Criteria:

* Unable to give valid informed consent
* Contraindications to MRI or MRI contrast agents
* A high risk factor for nephrogenic systemic fibrosis (NFS), including being on dialysis
* Suffering from heart disease, diabetes, single kidney, hypertension/hypotension, a history of renal disease, multiple myeloma, peripheral vascular disease
* Taking specific medications (loop diuretics, NSAIDs, aminoglycosides, vancomycin, amphotericin B or immunosuppressants)
* Claustrophobia
* Prior hormonal or radiation therapy for prostate cancer
* Active prostatitis, moderate to severe rectal inflammation, previous rectal surgery, or prostate biopsy within 12 weeks of planned MRI
* Currently or previously taking androgen deprivation therapy (however, use of a 5-α reductase inhibitor is allowed, provided it was discontinued at least 1 month prior to and 1 month following study entry)
* Have received, or are scheduled to receive, another IMP from 1 month prior to 1 month after inclusion in this study
* BMI of less than 18.5 or greater than 32
* Congestive heart failure, a past or present medical history of clinically significant electrocardiogram (EKG) abnormalities, which may include QT prolongation, a family history of prolonged QT interval syndrome, or a myocardial infarction (MI) within the past 12 months with ensuing unstable EKG, or ongoing acute or chronic pulmonary bronchospastic disease, including a history of chronic obstructive pulmonary disease or asthma, with an exacerbation within the past year

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Ability of the MRI machine to produce an image of the participant's prostate following an injection of Hyperpolarized Pyruvate (13C) as assessed by the physician | 2 years
  Feasibility of acquiring time resolved, 3D 13C lactate images from subjects with prostate cancer.

SECONDARY OUTCOMES:
Ability of the MRI machine to aid in predicting Gleason grade following an injection of Hyperpolarized Pyruvate (13C) as assessed by the physician | 2 years
  * Correlation between images obtained following Hyperpolarized Pyruvate (13C) Injection and the Gleason grade.
  * Added value for localizing clinically significant prostate carcinoma and predicting Gleason grade

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada